CLINICAL TRIAL: NCT00298857
Title: An Open-label, Prospective Trial to Determine the Effect(s) of Obesity on the Pharmacokinetic Parameters of Valproic Acid
Brief Title: A Pharmacokinetic Study to Compare the Dosing of Valproic Acid in Subjects With Different Body Weights
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05.02.045
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Healthy; Obesity; Pharmacokinetics
Keywords: Healthy; Obesity; Pharmacokinetics
MeSH Terms: conditions — Obesity | interventions — Valproic Acid

INTERVENTIONS:
Drug: Valproic acid

SUMMARY:
The purpose of this study is to compare the blood levels of valproic acid in subjects with different body weights and to evaluate whether the pharmacokinetic parameters of this drug is altered in the obese population.

DETAILED DESCRIPTION:
Many pharmacologic agents are dosed based on the weight of the patient, and studies are conducted to determine the appropriate doses of drugs for patients with different weights in order to find the safest and most effective dose for various weights. Valproic acid is a commonly used agent for the treatment of epilepsy, as well as migraine headaches and psychiatric disorders. This prospective study is designed to evaluate the effects of obesity on the pharmacokinetic parameters of valproic acid when compared to individuals at their healthy weight.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 21-60 years
* Normal healthy volunteers as per interview at screening
* Willing and able to provide written informed consent and comply with the study protocol

Exclusion Criteria:

* Inability to take oral medications
* pregnant or lactating females
* known hypersensitivity to valproic acid
* BMI less than 18.5 kg/m^2
* BMI between 25 and 29.9 kg/m^2, inclusive
* Taking any drug or dietary supplement within one week prior to study period
* Consumption of food 6 hours prior to study drug ingestion
* Know family history or history of urea cycle disorders
* Past history of pancreatitis
* Past history of liver disease

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2006-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve (AUC) from zero time to the 54-hour blood sampling and clearance in obese verses non-obese subjects after taking valproic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ettinger, MD, Principal Investigator — North Shore - Long Island Jewish Medical Center
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States